CLINICAL TRIAL: NCT03114020
Title: Phase 2 Randomized Parallel-Group Double-Blind Placebo-Controlled Multiple-Dose Proof-of-Concept Study to Evaluate the Efficacy/Safety of Hyaluronic Acid Inhalation Solution for Treatment of Emphysema
Brief Title: Efficacy/Safety of HA Inhalation Solution for Hereditary Emphysema in Patients With Alpha-1 Antitrypsin Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gerard Turino (Individual)
Responsible Party: Sponsor-Investigator, Gerard Turino, Sponsor-Investigator, Turino, Gerard, M.D.
Organization: Turino, Gerard, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C100-008
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Emphysema; Alpha 1-Antitrypsin Deficiency
Keywords: Emphysema; COPD; Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — Emphysema; alpha 1-Antitrypsin Deficiency; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: treatment has blinded labeling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hyaluronic Acid inhalation solution (Experimental): 3mL of 0.03% Hyaluronic Acid inhalation solution BID for 28 days
  Interventions: Drug: Hyaluronic Acid Inhalation Solution
- Placebo Inhalation Solution (Placebo Comparator): 3mL matching placebo inhalation solution BID for 28 days
  Interventions: Drug: Placebo Inhalation Solution

INTERVENTIONS:
Drug: Hyaluronic Acid Inhalation Solution — twice a day 3 mL of 0.03% Hyaluronic Acid Inhalation Solution
  Other Names: active inhalation solution
  Arms: Hyaluronic Acid inhalation solution
Drug: Placebo Inhalation Solution — Twice a day 3 ml of placebo inhalation solution
  Arms: Placebo Inhalation Solution

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of administering repeated doses of Hyaluronic Acid Inhalation Solution to subjects with Emphysema that have Alpha-1-Antitrypsin deficiency

DETAILED DESCRIPTION:
The study primarily aims to establish desmosine and isodesmosine concentrations in plasma, sputum and urine measured as markers of elastin degradation systemically in the lung and also markers of inflammation and fibrinogen. Assessment of vital signs, lab tests, carbon monoxide diffusing capacity, oxygen saturation, pulmonary function tests, ECGs, physical exams and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and comply with study requirements
2. Men or women aged 18 through 80 years at the time of consent
3. Diagnosis of emphysema at screening consistent with National Institutes of Health guidelines 19 GOLD COPD classification stages I, II or III
4. Evidence of emphysema on radiographic imaging.
5. A ratio of pre-bronchodilator FEV1 to forced vital capacity (FVC) of ≤ 80% at screening
6. FEV1 ≥ 30% and ≤ 79% (post-bronchodilator) of predicted normal at screening
7. Clinical laboratory tests (complete blood count, serum chemistry, and urinalysis) within normal limits or clinically acceptable to the PI and sponsor at screening
8. Women of childbearing potential and men who are sexually active must agree to use an adequate method of contraception (oral contraceptives, depot progesterone, condom plus spermicidal, or IUD) during the study and for 1 month after the final dose of study drug.
9. Evidence of alpha-1 antitrypsin deficiency (AATD) with any genotype except PiMZ deficiency. Individuals with PiMZ deficiency are not allowed in the study.
10. Patients must have stopped using Intravenous alpha-1 antitrypsin protein (AAT) augmentation therapy at least 3 months before entering study.

Exclusion Criteria:

1. Subjects with measured DLCO of ≤ 35%, or unable to perform a reproducible DLCO
2. Subjects unable to perform 3 reproducible spirometry tests after 8 attempts
3. Upper or lower respiratory tract infection within 2 weeks prior to screening and baseline (day1)
4. Presence of clinically relevant abnormality on chest x-ray (other than evidence of emphysema) within the previous 12 months
5. Use of supplemental oxygen therapy
6. Requirement for ventilator support within the last year
7. Exacerbation requiring treatment with systemic corticosteroids within the last 3 months
8. History of lung transplant or liver transplant.
9. Presence of clinically relevant abnormality on electrocardiogram (ECG)
10. Any medical condition that, in the investigator's judgment, would compromise study participation or the evaluation of the study drug
11. Women who are pregnant or breastfeeding
12. Receipt of an investigational drug within 30 days prior to screening
13. Patients who are current smokers or have smoked within the last 3 months -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Measurement of sputum, plasma and urine concentrations of desmosine and isodesmosine | 28 days
  measurement of biomarkers
Assessment of pulmonary function tests | 28 days
  measurement of pulmonary function

SECONDARY OUTCOMES:
Assessment of St. George Respiratory Questionnaire | 28 days
  measurement of patient abilities

CONTACTS AND LOCATIONS:
Overall Officials: Gerard M Turino, MD, Principal Investigator — Mount Sinai St Lukes
Locations (6):
- United States (5):
  - University of Miami Hospital, Miami, Florida
  - Pulmonary Health Physicians, PC, Fayetteville, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Science Center, Tyler, Texas
  - Medical College of Wisconsin / Froedtert Hospital, Milwaukee, Wisconsin
- Inspiration Research Limited, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No